CLINICAL TRIAL: NCT04640779
Title: Phase Ib Trial of Low-Dose Selinexor (KPT-330) in Combination With Choline Salicylate (CS) for the Treatment of Patients With Non-Hodgkin Lymphoma (NHL), Hodgkin Lymphoma, Histiocytic/Dendritic Cell Neoplasms, or Multiple Myeloma
Brief Title: Low-Dose Selinexor and Choline Salicylate for Non-Hodgkin or Hodgkin Lymphoma, Histiocytic/Dendritic Cell Neoplasm, or Relapsed or Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LS1981; P50CA097274 (NIH); NCI-2020-09704 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-009349 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2020-11-12; First posted 2020-11-23 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Histiocytic and Dendritic Cell Neoplasm; Recurrent Hodgkin Lymphoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Plasma Cell Myeloma; Refractory Histiocytic and Dendritic Cell Neoplasm; Refractory Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Multiple Myeloma | interventions — choline salicylate; selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (selinexor, choline salicylate) (Experimental): Patients receive selinexor PO BIW on days 1, 3, 8, 10, 15, 17, 22, and 24, and choline salicylate PO TID on days 1-28. Patients undergoing pharmacokinetic analysis receive choline salicylate beginning on D3C1 and beginning on day 1 of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patents who achieve >= stable disease continue treatment for an additional 6 cycles (maximum of 12 cycles) at the discretion of the treating physician and patient.
  Interventions: Drug: Choline Salicylate; Drug: Selinexor

INTERVENTIONS:
Drug: Choline Salicylate — Given PO
Drug: Selinexor — Given PO
  Other Names: ATG-010; CRM1 Nuclear Export Inhibitor KPT-330; KPT-330; Selective Inhibitor of Nuclear Export KPT-330; SINE KPT-330; Xpovio

SUMMARY:
This phase Ib trial evaluates the side effects and best dose of choline salicylate given together with a low dose of selinexor in treating patients with non-Hodgkin or Hodgkin lymphoma, or multiple myeloma whose prior treatment did not help their cancer (refractory) or for patients with histiocytic/dendritic cell neoplasm. Anti-inflammatory drugs, such as choline salicylate lower the body's immune response and are used with other drugs in the treatment of some types of cancer. Selinexor may stop the growth of cancer cells by blocking a protein called CRM1 that is needed for cell growth. This trial may help doctors learn more about selinexor and choline salicylate as a treatment for with non-Hodgkin or Hodgkin lymphoma, histiocytic/dendritic cell neoplasm, multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the maximum tolerated dose (MTD) of choline salicylate (CS) that can be combined with selinexor twice weekly in patients with relapsed/refractory non-Hodgkin, Hodgkin lymphoma, histiocytic/dendritic cell neoplasms, or relapsed/refractory (RR) multiple myeloma (MM).

SECONDARY OBJECTIVE:

I. To evaluate the response [overall response rate (ORR), clinical benefit rate (CBR) and duration of response (DOR)) of selinexor and CS in patients with relapsed/refractory non-Hodgkin or Hodgkin lymphoma, histiocytic/dendritic cell neoplasms, or multiple myeloma.

CORRELATIVE RESEARCH OBJECTIVE:

I. To determine if CRM1, RAD51, gH2AX, BRCA1 and 53BP1 expressions in malignant lymphoma cells, extramedullary myeloma, or histiocytic/dendritic cell neoplasm cells from those patients treated on this study have a predictive role.

OUTLINE: This is a dose-escalation study.

Patients receive selinexor orally (PO) twice a week (BIW) on days 1, 3, 8, 10, 15, 17, 22, and 24, and choline salicylate PO three times daily (TID) on days 1-28. Patients undergoing pharmacokinetic analysis receive choline salicylate beginning on day 3 of cycle 1 (D3C1) and beginning on day 1 of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patents who achieve >= stable disease continue treatment for an additional 6 cycles (maximum of 12 cycles) at the discretion of the treating physician and patient.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Non Hodgkin or Hodgkin lymphoma or histiocytic/dendritic cell neoplasm meeting one of the following criteria:

  * Biopsy-proven relapsed and/or refractory Non-Hodgkin or Hodgkin lymphoma or histiocytic/dendritic cell neoplasms

    * Relapsed is defined as a relapse that occurred after having a response to the last therapy that lasted > 26 weeks
    * Refractory is no response (stable disease or progressive disease while on therapy) or relapse within 6 months. Refractoriness to autologous stem cell transplant will be defined as disease progression within 52 weeks following transplant OR

Multiple myeloma neoplasm meeting the following criteria:

* Relapsed and/or refractory multiple myeloma (RRMM) as per the International Myeloma Working Group (IMWG) uniform criteria
* If extramedullary myeloma, most recent tumor biopsy must be < 26 weeks prior to registration

  * Measurable or assessable disease:
* For Non-Hodgkin or Hodgkin Lymphoma and histiocytic/dendritic cell:

  * Measurable disease is defined as measurable by computed tomography (CT) [dedicated CT or the CT portion of a positron emission tomography (PET)/CT] or MRI: To be considered measurable, there must be at least one lesion that has a single diameter of >= 1.5 cm NOTE: Skin lesions can be used if the area is >= 1.5 cm in at least one diameter and photographed with a ruler. Patients with assessable disease by PET/CT are also eligible as long as the assessable disease is biopsy proven lymphoma or histiocytic/dendritic cell neoplasms
* For Multiple myeloma:
* Measurable disease by IMWG criteria as defined by at least one of the following:

  * Serum M-protein >= 0.5 g/dL
  * Urine M-protein >= 200 mg in a 24-hour collection
  * Serum Free Light Chain level >= 10 mg/dL provided the free light chain ratio is abnormal
  * Measurable plasmacytoma (at least one lesion that has a single diameter of >= 2 cm on CT portion of PET/CT scan or MRI)
  * Bone marrow plasma cells >= 10%

    * Exception: A patient with non-secretory multiple myeloma (MM) but with bone marrow plasma cells >= 30% may be considered for enrollment after discussion with the PI that includes the feasibility of an individualized plan for response assessment
  * Patients with Immunoglobulin A (IgA) or Immunoglobulin D (IgD) myeloma in whom serum protein electrophoresis is deemed unreliable, due to co-migration of normal serum proteins with the para protein in the beta region, may be considered eligible as long as total serum IgA or IgD level is elevated above normal range

    * Patients with non-Hodgkin or Hodgkin lymphoma must have previously been treated with >= 2 lines of therapy
    * Patients with histiocytic/dendritic cell neoplasms must previously have been treated with >= 1 line of therapy
    * Patients with RRMM must have received ≥4 prior therapies whose disease is refractory to >= 2 proteasome inhibitors, >= 2 immunomodulatory agents, and an anti-CD38 monoclonal antibody
    * Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2
    * Absolute neutrophil count (ANC) >= 1,000/mm^3 (obtained =< 14 days prior to registration)
    * Platelet count >= 100,000/mm^3 (obtained =< 14 days prior to registration)
    * Hemoglobin >= 8.5 g/dL (may be transfused to reach criteria) (obtained =< 14 days prior to registration)
    * Total bilirubin < 2 x upper limit of normal (ULN) (or total bilirubin =< 3.0 x ULN with direct bilirubin =< 1.5 x ULN in patients with well-documented Gilbert's syndrome) (obtained =< 14 days prior to registration)
    * Aspartate transaminase (AST) =< 2.5 x ULN and alanine aminotransferase (ALT) =< 2.5 x ULN (obtained =< 14 days prior to registration)
    * Calculated creatinine clearance must be >= 35 ml/min using the Cockcroft Gault formula (obtained =< 14 days prior to registration)
    * Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
    * Female of childbearing potential (FCBP*) must commit to take highly effective contraceptive precautions** without interruption during the study and continue for at least 12 weeks after the last dose of selinexor and CS. FCBP must refrain from breastfeeding and donating oocytes during the course of the study. Males must use an effective barrier method of contraception without interruption during the study and continue for at least 12 weeks after the last dose of selinexor and CS. They must refrain from donating sperm during the study participation.
* *FCBP defined as sexually mature women who have not undergone bilateral tubal ligation, bilateral oophorectomy, or hysterectomy; or who have not been postmenopausal (i.e., who have not menstruated at all) for at least 1 year

  * Highly effective forms of birth control are methods that achieve a failure rate of less than 1% per year when used consistently and correctly. Highly effective forms of birth control include: hormonal contraceptives (oral, injectable, patch, and intrauterine devices), male partner sterilization, or total abstinence from heterosexual intercourse, when this is the preferred and usual lifestyle of the patient NOTE: The double-barrier method (e.g., synthetic condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel), periodic abstinence (such as calendar, symptothermal, post-ovulation), withdrawal (coitus interruptus), lactational amenorrhea method, and spermicide-only are not acceptable as highly effective methods of contraception

    * Provide written informed consent
    * Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
    * Willingness to provide mandatory blood specimens per protocol for Pharmacokinetics (PKs) and banking
    * For lymphoma, extramedullary myeloma and histiocytic/dendritic cell neoplasms, willing to provide mandatory tissue samples for correlative research. NOTE: If an institution is not able to provide the tissue, it does not cause the patient to be ineligible; however, the collection of these tissues is strongly recommended.

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Patients known to have active hepatitis B, or C infection, or known to be positive for hepatitis C virus (HCV) ribonucleic acid (RNA) or hepatitis B surface antigen (HBsAg) [hepatitis B virus (HBV) surface antigen]. Patients known to be human immunodeficiency virus (HIV) positive, except those with CD4+ T-cell (CD4+) counts >= 350 cells/microliter (µL) and on an established antiretroviral therapy (ART) for at least twelve weeks and have an HIV viral load less than 400 copies/mL prior to enrollment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Life expectancy of < 6 months
* Active gastrointestinal (GI) dysfunction interfering with the ability to swallow tablets, or any GI dysfunction that could interfere with absorption of study treatment
* Known intolerance to or contraindications for choline salicylate therapy. Patients with known allergy to acetylsalicylic acid (ASA) are not eligible
* Prior exposure to a selective inhibitors of nuclear export (SINE) compound, including selinexor
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Active second malignancy requiring treatment that would interfere with the assessment of the response of the primary cancer to this protocol therapy. Patients with treated malignancies on hormonal therapy (for example breast or prostate cancer) are eligible
* History of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Radiation, chemotherapy, or immunotherapy or any other anticancer therapy =< 2 weeks prior to registration. NOTE: Exception: patients on any Bruton tyrosine kinase (BTK) inhibitor (ibrutinib, zanabrutinib, acalabrutinib, etc), or venetoclax, or corticosteroids (any dose) may continue therapy up until the new regimen has started at investigator discretion. After the start of protocol therapy, corticosteroids can be used at investigator's discretion and tapered to lowest possible dose
* Active graft versus (vs.) host disease (after allogeneic stem cell transplantation) at registration
* Major surgery (including bowel resection) =< 3 weeks prior to registration
* Must not be currently eligible or have declined high-dose therapy with autologous stem cell transplantation rescue or chimeric antigen receptor (CAR)-T cell therapy
* Primary mediastinal (thymic) large B-cell lymphoma (PMBL)
* Known active central nervous system (CNS) lymphoma. Patients with previous CNS involvement can enroll if the CNS component is inactive
* Patients who are on active anticoagulant therapy with direct oral anticoagulants (DOACs), aspirin or warfarin are not eligible due to potential bleeding. EXCEPTIONS: Patients who are on aspirin (81 mg) for primary prevention of cardiovascular disease can enroll, but the ASA needs to be held while on this protocol therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of the combination of low-dose selinexor with choline salicylate | Up to 12 cycles (a cycle is 28 days)
  Defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients (at least 2 of a maximum of 6 new patients).

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 12 cycles
  Adverse events will be assessed according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns (overall and by dose level). Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.
Overall response rate | Up to 12 cycles (a cycle is 28 days)
  Noted as the objective status at any time before progression or initiation of new treatment. Response will be evaluated using all cycles of treatment. Defined as the following for patients with Multiple Myeloma: stringent Complete Response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), minimal response (MR), stable disease (SD), progressive disease (PD), and clinical relapse (REL). Defined as the following for patients with Non-Hodgkin or Hodgkin lymphoma or Histiocytic/dendritic cell neoplasms: complete metabolic response (CMR), partial metabolic response (PMR), or prolonged stable disease (SD) (duration of at least 3 months).
Clinical benefit rate | Up to 12 cycles (a cycle is 28 days)
  Noted as the objective status at any time before progression or initiation of new treatment. Response will be evaluated using all cycles of treatment. Defined as the following for patients with Multiple Myeloma: sCR, CR, VGPR, PR, MR, SD, PD, and REL. Defined as the following for patients with Non-Hodgkin or Hodgkin lymphoma or Histiocytic/dendritic cell neoplasms: CMR, PMR, or prolonged SD (duration of at least 3 months).
Duration of response | Up to 12 cycles (a cycle is 28 days)
  Defined for all evaluable patients who have achieved a response as the date at which the patient's objective status is first noted to the earliest date progression is documented.

OTHER OUTCOMES:
CRM1 expression | Up to 12 cycles (a cycle is 28 days)
  Will determine if the CRM1 expression grade, via immunohistochemistry and reported as grade 1 (low), grade 2 (moderate) and grade 3 (high), in malignant cells correlates with overall response rate after treatment with selinexor.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Paludo, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2025-09-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT04640779/ICF_000.pdf